CLINICAL TRIAL: NCT05539924
Title: A Comparison Between Pregabalin and Gabapentin as Adjuvants to Opioids in Elective Lumber Micro Discectomy to Control Postoperative Pain. (A Prospective Randomized Controlled Study)
Brief Title: Pregabalin Versus Gabapentin Opioid Sparing Effect in Discectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00arafa00
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Opioid Use
MeSH Terms: interventions — Pregabalin; Gabapentin; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group P (Active Comparator): The patients in this group will receive 150 mg pregabalin tablets P.O 1 hours before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.
  Interventions: Drug: Pregabalin 150mg gabapentin 400mg
- Group G (Active Comparator): The patients in this group will receive 400 mg Gababentin4 tablets P.O 1 hours before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.
  Interventions: Drug: Pregabalin 150mg gabapentin 400mg
- Group C (Placebo Comparator): The patients in this group will receive vitamin B12 (100µg) as placebo tablets P.O hours before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.
  Interventions: Drug: Pregabalin 150mg gabapentin 400mg

INTERVENTIONS:
Drug: Pregabalin 150mg gabapentin 400mg — oral administration
  Other Names: vitamin B12

SUMMARY:
Pregabalin and gabapentin are both GABA analogue and their mechanism of action is not fully understood. Both drugs when given as a pre-emptive analgesia for spinal surgery were found to reduce intra-and postoperative opioid requirements.

Preoperative intramuscular injection of morphine could reduce the patients' pain during the percutaneous transformational endoscopic discectomy "PTED" surgery and improve the patients' satisfaction without affecting the surgical outcome. The efficacy of adding pregabalin or gabapentin to preoperative intramuscular morphine is not yet investigated.

The current study aims to compare the analgesic effect of both drugs when given preoperatively with intramuscular morphine.

DETAILED DESCRIPTION:
Preoperative assessment will be conducted on the patients that will be enrolled in this study including history taking, Physical examination, and laboratory investigations and radiological investigations; according to the medical condition of the patients. All patients must fulfill the inclusion criteria then the patients are consented to be included in the study & informed about the required fasting hours.

Informed consent will be obtained from the entire patient enrolled in this study on the day before surgery. VAS score will be explained to all the patients' Visual analogue scale to measure post-operative pain.

VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end.

The patient marks on the line the point that they feel represents their perception of their current state. On the day of surgery, study drug was given orally 1 hour before the time of induction of anesthesia.

In the operation theatre, baseline heart rate, oxygen saturation, and mean arterial blood pressure were recorded. After insertion of a wide bore cannula, and premeditations will be given including anxiolytics e.g. midazolam (70-80mcg/kg) not to exceed >5mg and Ondansteron (4mg)

Then the patients will be randomized into one of the following three groups:

Group P: The patients in this group will receive 150 mg pregabalin tablets P.O 1 hour before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.

Group G: The patients in this group will receive 400 mg Gababentin4 tablets P.O 1 hour before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.

Group C: The patients in this group will receive vitamin B12(100µg) as placebo tablets P.O 1 hour before surgery then after half hour morphine 0.1 mg/kg will be administered intramuscularly.

The patients enrolled in the study will be transferred to Operation room and monitored all through the surgical procedure using pulse oximeter, non-invasive blood pressure, ECG, capnogram. Patient will be preoxygenated with 100% oxygen for 3 minutes prior to induction. Induction of Anaesthesia will be done using propofol (2mg/kg), Fentanyl (1mcg/kg) and Atracrium (0.5 mg/kg) then Endotracheal intubation will be inserted smoothly using Oral ETT (ID 7.5mm in adult male and ID 7 mm in adult female) then position of Endotracheal tube will be confirmed with auscultation and Capnography.

Anaesthesia will be maintained using 1.2 % isoflurane (that will be adjusted according to hemodynamics changes) with top up doses of atracurium (0.1 mg/kg) every 30 minutes.

Ventilation will be maintained using volume controlled mode with the following parameters:

Tidal volumes 6-8 ml/kg, Respiratory Rate 12 breath/minute to achieve end tidal CO2 between 30 to 35 mmHg.

Intraoperative hemodynamics including heart rate, blood pressure (Systolic, Diastolic and Mean Arterial pressure) will be measured as baseline before induction, after ¼ hour from intubation, before and after the patient being in prone position and every ½ hour.

The patient will be positioned in prone position and precautions of this position will be applied, if Intraoperative hemodynamic changes happened more than 20% or 25% from baseline hemodynamic readings due to lack of analgesia, we will administer(0.5-1 mic.) Fentanyl as rescue analgesia.

At the End of the operation the patient will be returned to supine position and awaked fully reversed with injection of neostigmine and Atropine, and the patients will be extubated and shifted to Recovery room and we will check hemodynamics including heart rate and systolic, diastolic, mean arterial blood pressure, assess VAS scale and requirement of rescue analgesia (morphine) in zero hour then the patients will be transferred to the ward and reassess hemodynamics, the VAS scale and requirement of rescue analgesia after two hours, four hours, six hours, eight hours, ten hours, twelve hours, sixteen hours, twenty hours and twenty four hours respectively.

Postoperative pain assessment through VAS will be according to the scale as follow:

* Pain level 0: no pain
* Pain level1-3: mild pain
* Pain level 4-6: moderate pain
* Pain level 7-10: severe pain

  1. Postoperative pain will be managed as follow:
* Mild pain will be treated with paracetamol 1 gm. IV.
* Moderate pain will be treated with paracetamol 1 gm. IV & ketolac 30 mg IV.
* Severe pain will be treated with morphine 3mg (rescue analgesia). Then patient will be reassessed and recorded as mentioned above and the specific treatment will be repeated after 8 hours from the initial dose according to VAS.

  2. Opioids complications such as respiratory depression will be recorded and managed supportively by oxygen mask, controlled airway and if persistent or severe hypoventilation occurs positive pressure ventilation may be needed, nausea and vomiting will be treated with ondansterone (4 mg IV).

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II

  * Elective Lumber micro discectomy.
  * BMI ≤ 35
  * Time of operation not exceeding 2hours.

Exclusion Criteria:

* Patients' refusal

  * Age < 20 years or > 60 years
  * ASA III to ASA IV
  * Contraindications to Opioids e.g., Allergy, Bronchial asthma.
  * Contraindication to Pregabalin or Gabapentin e.g. Allergy
  * Psychological or mental disorders.
  * Disturbance of Conscious level.
  * Uncooperative patients.
  * Patients with impaired renal function or creatinine clearance less than 50ml/min

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesia during the first postoperative 24 hours. | 24 hours
  call for analgesia

SECONDARY OUTCOMES:
pain score | 24 hours post operative
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: mohamed s arafa, MD, Study Director — kasr el aini H
Locations (1):
- kasr el aini H, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No